CLINICAL TRIAL: NCT07178067
Title: Short Chain Fatty Acids Profiles in Amyotrophic Lateral Sclerosis: Longitudinal Effects of Disease and Mediterranean Diet Intervention
Brief Title: Longitudinal Evaluation of Short-Chain Fatty Acid Profiles During the Natural Disease Course and a Mediterranean Diet Intervention in Amyotrophic Lateral Sclerosis Patients
Acronym: IMPACT-ALS
Status: Completed | Type: Observational
Sponsor: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other)
Responsible Party: Principal Investigator, Motataianu Anca, Associate Professor, George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures
Other Study IDs: TE 74/2022; PN-III-P1-1.1-TE-2021-0960 (Other Grant/Funding Number: The Ministry of Research, Innovation, and Digitization, CNCS-UEFISCDI)
Record Dates: First submitted 2025-09-03; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: short-chain fatty acid; amyotrophic lateral sclerosis; microbiota-gut-brain axis; LC-MS/MS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Diet, Mediterranean

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALS patients: 44 patients diagnosed with amyotrophic lateral sclerosis (ALS) in the past 12 months.
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Mediterranean diet — The Mediterranean diet, characterised by a high intake of fruits, vegetables, whole grains, legumes, nuts, and olive oil, along with moderate consumption of fish and poultry, has been associated with anti-inflammatory and neuroprotective effects. Notably, this dietary pattern has the potential to enhance the production of short-chain fatty acids (SCFAs) and support gut microbial diversity, representing a promising strategy for nutritional intervention in patients with ALS.

SUMMARY:
This observational study explored the connection between the gut microbiota and the brain in patients with amyotrophic lateral sclerosis (ALS), specifically the modulation of short-chain fatty acids during disease progression and after following a Mediterranean diet for 6 months. Recent research suggests that the gut microbiome-the community of bacteria and other microorganisms living in our intestines-may influence how ALS develops and progresses. The hypothesis was that changes in the gut microbiome and the substances it produces, such as short-chain fatty acids (SCFAs), may play an important role in ALS progression. Additionally, the effect of the Mediterranean diet on circulating short-chain fatty acid concentrations was assessed.

DETAILED DESCRIPTION:
This study investigates the role of the microbiome-gut-brain axis in the progression of amyotrophic lateral sclerosis (ALS), with a focus on short-chain fatty acids (SCFAs) and their associated biomarker panel (SCFAGGYC-PROF). The investigators hypothesized that alterations in the gut microbiota composition and SCFA metabolism contribute to the heterogeneity of ALS phenotypes, influencing whether the disease follows a rapidly progressive or more slowly progressive course.

Participants with ALS and healthy controls undergo blood sampling and stool collection at baseline and follow-up. Serum analyses include: measurement of circulating SCFA levels using liquid chromatography-tandem mass spectrometry (LC-MS/MS).

In a subset of ALS patients, dietary interventions consistent with a Mediterranean dietary pattern are introduced to evaluate the impact of nutrition on gut microbiota composition, SCFA production, and clinical disease progression. This 12-month study (6 months natural course + 6 months dietary intervention) evaluated Mediterranean diet effects on ALS progression rate and circulating levels of SCFA. The diet-known for neuroprotective and anti-inflammatory properties-was associated with significant changes in SCFA plasma levels.

A key process stage involved developing and applying an LC-MS/MS method for plasma quantification of acetic (C2), propionic (C3), butyric (C4), 3-hydroxybutyric (3-OH-C4), hexanoic (C6), and iso-hexanoic acid (Iso-C6; 4-methyl-valeric), using acetic acid-C13, butyric-d8 and hexanoic-d11 as internal standards.

After extraction and derivatization of analytes from plasma, samples were analyzed by reversed-phase LC and detected via MS/MS in MRM mode with negative ESI. The method enabled quantitative determination of free plasma carboxylic acids.

Analytical development and performance verification were carried out for simultaneous analysis of 6 short-chain carboxylic acids plus 3 homologous internal standards via LC-MS/MS with prior derivatization using EDC, 3-NPH, and pyridine. Validation covered LOD/LOQ, linear range and signal-concentration dependence (R>0.9900), accuracy (85-115%), inter-series precision (<15%), and carryover (none), ensuring confidence in the method.

Working solutions were prepared from STOCK/STD solutions fresh each day for method/derivatization checks and for spiking blank plasma at defined levels to build daily calibration curves for routine analysis. Solvent water:methanol 3:7 (v/v) was freshly prepared each analysis day.

Samples were prepared fresh on analysis day and immediately loaded in the autosampler. Samples were grouped into 4 batches: Control, T0, T1, T2. Plasmas were thawed once and equilibrated to room temperature. Sample preparation mirrored that of calibration/control plasma, spiked only with internal standards.

Quantification of SCFAs in Control (n=40), T0 (n=44), T1 (n=36), T2 (n=30). Each batch was run independently with fresh daily calibration curves from pooled healthy plasma spiked at method concentrations. Blanks (unspiked plasma and ISTD-only plasma) were also run to assess endogenous signal. Curves were 6-point linear (R>0.9900), used for quantification with internal-standard peak area correction: acetate C2, propionate C3, and 3-OH-C4 with acetate-C13 ISTD; butyrate C4 with butyrate-d8 ISTD; iso-hexanoic (Iso-C6) and hexanoic C6 with hexanoic-d11 ISTD.

Statistical interpretation using descriptive statistics per analyte and batch: means, SD, %CV (RSD), min, max. Chromatographic peaks processed in MultiQuant (Sciex) linked to Analyst 1.7.1; data/statistics in Microsoft Excel 2019. Method validated for sensitivity, selectivity, linearity, LLOQ, carryover, within-run/between-run precision and accuracy, and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with amyotrophic lateral sclerosis (ALS) in the past 12 months.
* Disease duration of less than 1 year.
* Fulfillment of the El Escorial diagnostic criteria (1996) for clinically probable or clinically definite ALS.

Exclusion Criteria:

* Patients with an expected survival <18 months.
* Presence of other neurodegenerative diseases.
* Major comorbidities, such as: heart failure, cancer, autoimmune diseases, systemic diseases.
* Gastrointestinal diseases that could influence gut microbiota.
* Recent or ongoing treatment with antibiotics, probiotics, or prebiotics.
* Low compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective, single-center study enrolled adults from Romania diagnosed with ALS at Neurology Clinic 1, Mureș County Clinical Emergency Hospital , with an ALS diagnosis within the past 12 months, disease duration under 1 year, El Escorial (1996) criteria-clinically probable or clinically definite ALS. ALS cohort: N=44 at baseline (T0, Aug-Oct 2022); mean age 58.4 ± 12.5 years; 28 men / 16 women. Follow-up: T1 (6 months): N=36 (8 deaths by T1). T2 (12 months): N=30 (6 additional deaths between T1 and T2). Healthy controls: N=40, age- and sex-matched community volunteers without known neurodegenerative or major systemic disease. The patients were recruited through consecutive recruitment at the Neurology Clinic 1, Mureș County Clinical Emergency Hospital (Târgu Mureș, Romania) over a 3-month window (01 Aug-31 Oct 2022).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Analysis of serum SCFA levels in ALS patients and healthy controls, and evaluating the change in circulating SCFA concentrations associated with Mediterranean diet intervention | 12 months
  This study compares plasma levels of short-chain fatty acids (SCFAs): acetic acid (ng/mL), propanoic acid (ng/mL), butyric acid (ng/mL), 3-OH butyric acid, 4-methyl-valeric acid (ng/mL) between adults with amyotrophic lateral sclerosis (ALS) and age/sex-matched healthy controls at baseline (T0) and then tracks how these levels change after 6 months of natural disease progression (T1) and 6 months after introducing a Mediterranean diet (T2) in ALS patients. Outcomes: Mean SCFA concentrations (±SD) (ng/mL) at T0 between-group (ALS vs control) differences at baseline, and within-patient changes over time to assess whether the Mediterranean diet is associated with favorable SCFA shifts (T0-T1, T1-T2).

SECONDARY OUTCOMES:
Association of Serum SCFA Levels With ALS Progression Measured by ALSFRS-R at T0, T1, and T2 | 12 months
  The investigators analysed whether mean plasma levels of short-chain fatty acids (SCFAs)-acetate, propionate, butyrate, 3-hydroxybutyrate, hexanoate, and iso-hexanoate (ng/mL)-are associated with clinical progression of amyotrophic lateral sclerosis (ALS) (ALSFRS-R progression rate (ΔPR).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine, Pharmacy, Science and Technology of Târgu Mureș 'George Emil Palade', Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: No
Given the small, regionally identifiable ALS cohort and the rarity of the condition, the risk of re-identification remains high even after de-identification.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT07178067/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT07178067/ICF_001.pdf